CLINICAL TRIAL: NCT05839639
Title: A Multicenter, Randomized, Controlled Phase IIa Study to Evaluate the Antiviral Activity and Safety of HH-003 Injection in Subjects With HBeAg-Negative Chronic Hepatitis B Treated With Nucleos(t)Ide Reverse Transcriptase Inhibitors
Brief Title: A Study to Evaluate the Antiviral Activity and Safety of HH-003 Injection in Subjects With HBeAg-Negative Chronic Hepatitis B Treated With Nucleos(t)Ide Reverse Transcriptase Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huahui Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HH003-202
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NrtIs (Active Comparator)
  Interventions: Drug: NrtIs
- HH-003 (Experimental)
  Interventions: Drug: HH-003
- HH-003+NrtIs (Experimental)
  Interventions: Drug: HH-003+NrtIs

INTERVENTIONS:
Drug: NrtIs — Subjects will receive NrtIs therapy for 24 weeks.
  Arms: NrtIs
Drug: HH-003 — Subjects will receive HH-003 20 mg/kg intravenously Q2W for 24 weeks.
  Arms: HH-003
Drug: HH-003+NrtIs — Subjects will receive HH-003 20 mg/kg intravenously Q2W for 24 weeks. Subjects will receive NrtIs therapy for 24 weeks.
  Arms: HH-003+NrtIs

SUMMARY:
This is a multicenter, randomized, controlled Phase IIa study of HH-003 injection, HH-003 injection is a monoclonal antibody targeting Hepatitis B virus. This study aims to evaluate the antiviral activity and safety in subjects with with HBeAg-negative Chronic Hepatitis B treated with nucleos(t)ide reverse transcriptase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Male or female aged from 18 to 65years (inclusively);
* 18 kg/m^2≤BMI≤32 kg/m^2, body weight≥45 kg for men and ≥40 kg for women;
* At screening, etiological, clinical, or pathological evidence indicates chronic hepatitis B virus infection for at least 6 months; and negative HBeAg for more than 6 months; 10 IU/mL≤HBsAg≤3000 IU/mL; HBV DNA≤20 IU/mL; ALT≤1×ULN;
* Participants who have been on the treatment of nucleos(t)ide reverse transcriptase inhibitors (limited to entecavir [ETV], tenofovir disoproxil fumarate [TDF], or tenofovir alafenamide fumarate [TAF]) for at least 3 years (as judged by the investigator) at screening.

Exclusion Criteria:

* Females who are pregnant or lactating at screening;
* History of alcoholic liver disease, non-alcoholic steatohepatitis, autoimmune liver disease, other hereditary liver disease, drug-induced liver disease or other clinically significant chronic liver disease induced by non-HBV infection;
* History or presence of progressive liver fibrosis or cirrhosis, including but not limited to liver stiffness measurement [LSM] ≥ 9 kPa at screening, progressive liver fibrosis or cirrhosis (e.g., S ≥ 3 in GS score or METAVIR ≥ F3) by liver histopathology examination, according to the Consensus on the diagnosis and therapy of hepatic fibrosis [2019]; or the presence of ascites, hepatic encephalopathy, upper gastrointestinal bleeding, or esophageal and gastric varices.
* History or presence of hepatocellular carcinoma, or alpha-fetoprotein (AFP) ≥ 50 ng/mL at screening; or suspicion of hepatocellular carcinoma indicated by liver ultrasound, CT, or MRI.
* Use of antiviral therapy with interferon within 1 year prior to screening
* Any of the following lab test results at screening: total bilirubin >2xULN or direct bilirubin >1.5xULN, hemoglobin <120 g/L for males or <110 g/L ro females, platelets count<100,000/mm^3 (100×10^9/L), and absolute neutrophils count <1,500/mm^3 (1.5×10^9/L), Serum albumin < 35 g/L; international normalized ratio (INR) of prothrombin time > 1.3; or estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-10-09 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving sustained viral response | From baseline to Week 24
Changes from baseline in serum HBsAg levels | From treatment start to Week 24

SECONDARY OUTCOMES:
Proportion of participants with undetectable HBV DNA in those with positive HBV DNA at baseline | From treatment start to Week 24
Proportion of participants achieving sustained viral response | From baseline to Week 48
Duration of sustained viral response | From treatment start to Week 48
Changes from baseline in serum HBsAg levels | From treatment start up to Week 48
Proportion of participants with HBV pgRNA negativation in those with positive HBV pgRNA at baseline | From baseline to Week 24
Proportion of participants with normal ALT levels | From treatment start to Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China